CLINICAL TRIAL: NCT03185520
Title: Longitudinal Study of Young Patients With Embolic Stroke of Undetermined Source (ESUS)
Brief Title: Young ESUS Patient Registry
Acronym: Y-ESUS
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Young ESUS
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: Stroke; Ischemic Stroke; Cryptogenic Stroke; Embolic stroke of undetermined source; ESUS; Cerebrovascular Disease
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to determine the clinical characteristics of young ESUS patients using diagnostic criteria of the Cryptogenic Stroke / ESUS International Working Group, and to determine the rates of stroke recurrence, death, and hospital readmission in a contemporary cohort of young ESUS patients during follow-up of up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Embolic stroke of undetermined source (ESUS) within 60 days, defined as:

   1. Recent ESUS (including transient ischemic attack with positive neuroimaging) visualized by brain computed tomography (CT) or magnetic resonance imaging (MRI) that is not lacunar (i.e., lacunar infarcts are subcortical infarcts ≤ 1.5 cm in the territory of middle cerebral artery or pons; infarcts involving the cerebellum or lateral medulla are not considered as lacunar infarcts). Patients with multiple simultaneous acute lacunar infarcts on diffusion weighted imaging may be included. In case of embolic large artery occlusions clearly documented on angiography who undergo successful recanalization, visualization of infarct on neuroimaging is not mandated, and
   2. Absence of cervical carotid atherosclerotic stenosis (or vertebral and basilar atherosclerotic stenosis in case of posterior circulation stroke), that is >50%, or occlusion in arteries supplying the area of ischemia, (unless deemed embolic) in CT or magnetic resonance (MR) angiography or conventional angiography or ultrasound, and
   3. No history of atrial fibrillation (AF), no documented AF on 12-lead electrocardiogram or episode of AF lasting 6 minutes or longer detected after ≥ 24-hour cardiac rhythm monitoring (Holter or telemetry; at least 20 hours acceptable), and
   4. No intra-cardiac thrombus on either transesophageal or transthoracic echocardiography, and
   5. No other specific cause of stroke identified by routine clinical care (e.g., arteritis, dissection, migraine/vasospasm, drug abuse)
2. Age ≥ 21 to ≤ 50 years
3. Written informed consent with local regulations governing research in human subjects

Exclusion Criteria:

1. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g., employee or student of the investigational site)
2. Enrollment in an investigational study on ESUS
3. If imaging of intracranial arteries are performed by CT or MR angiography, digital subtraction angiography or transcranial Doppler: >50% luminal stenosis or occlusion in arteries supplying the area of ischemia (unless deemed embolic)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presenting to hospital-based stroke unit with an ESUS Stroke
Sampling Method: Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Recurrent ischemic stroke and/or death in a well-defined Young ESUS cohort | Approximately 18 Months

SECONDARY OUTCOMES:
Recurrent ischemic stroke in a well-defined Young ESUS cohort | Approximately 18 Months
Prevalence of Patent Foramen Ovale in a well-defined Young ESUS cohort | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kanjana S Perera, MD, FRCPC, Principal Investigator — McMaster University, Hamilton Health Sciences, and Population Health Research Institute; Robert G Hart, MD, Principal Investigator — McMaster University and Population Health Research Institute
Locations (44):
- United States (7):
  - Stanford University, Stanford, California
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of South Carolina - School of Medicine - Neurology, Columbia, South Carolina
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - University of Texas Health Center - San Antonio, San Antonio, Texas
- Argentina (2):
  - Fundacion para la Lucha vs. Enf. Neurologicas de la Infancia, Buenos Aires, Buenos Aires
  - Complejo Médico de la PFA Churruca Visca, Buenos Aires, Buenos Aires
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Western Health, Footscray, Victoria
- Canada (6):
  - University of Calgary/Foothills Medical Center, Calgary, Alberta
  - Vancouver Stroke Program - Research Offices at Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital (Civic Campus), Ottawa, Ontario
  - University Health Network, Toronto, Ontario
- Clínica Alemana de Santiago, Santiago, Chile
- France (2):
  - Hopital Bichat, Paris
  - Versailles Hospital, Versailles
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Neurologische UNiversitätsklinik Erlangen, Erlangen
  - Asklepios Klinik Nord, Department of Neurology, Hamburg
- National Institute of Neurology and Neurosurgery, Mexico City, Mexico
- Poland (2):
  - Institute Psychiatry and Neurology, 2 Department of Neurology, Warsaw
  - Szpital Specjalistyczny im. Sw. Lukasza, Oddzial Neurologii z Oddzialem Udarowym, Gmina Końskie, Świętokrzyskie Voivodeship
- Tiervlei Trial Centre, Bellville, South Africa
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de La Santa Creu Isant Pau, Barcelona
  - Hospital Clínico Universitario, Valladolid
- Stroke Center Inselspital University Hospital Bern, Bern, Switzerland
- United Kingdom (13):
  - Buckinghamshire Healthcare NHS Trust, High Wycombe, Buckinghamshire
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - West Hertfordshire Hospitals NHS Trust, Watford, Hertfordshire
  - East Kent Hospitals - Queen Elizabeth the Queen Mother Hospital, Margate, Kent
  - Northwick Park Hospital, Harrow, Middlesex
  - Yoevil District Hospital Foundation Trust, Yeovil, Somerset
  - Cambridge University Foundation Trust Hospitals, Addenbrookes site, Cambridge
  - Gloucestershire Royal Hospital, Gloucester
  - Imperial College Healthcare NHS Trust, London
  - Royal Hallamshire Hospital, Sheffield
  - Southend University Hospital NHS Foundation Trust, Southend-on-Sea
  - Royal Stoke University Hospital, University Hospital of North Midlands NHS Trust, Stoke-on-Trent
  - Royal Wolverhampton Hospitals NHS trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No